CLINICAL TRIAL: NCT00764374
Title: A Long-term, Open-label, Uncontrolled Trial of YM443 (Z-338) in Patients With Functional Dyspepsia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 443-CL-501
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Dyspepsia; Functional Dyspepsia
Keywords: YM443; Z-338; Acotiamide; Rome III; Signs and symptoms, digestive
MeSH Terms: conditions — Dyspepsia; Signs and Symptoms, Digestive | interventions — Z 338

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: YM443

INTERVENTIONS:
Drug: YM443 — oral
  Other Names: Z-338; acotiamide

SUMMARY:
To examine the safety and efficacy of Z-338 (YM443) after long-term administration in patients with functional dyspepsia, and also to examine the pattern of long-term administration.

ELIGIBILITY:
Inclusion Criteria:

* Patient showing at least one of the following 4 symptoms from more than 6 months before obtaining consent

  * postprandial fullness
  * early satiation
  * upper abdominal pain
  * upper abdominal discomfort
* Patient showing at least 2 of the 8 symptoms shown below repeatedly from 3 months before obtaining consent (At least one symptom of either postprandial fullness or early satiation should be included.)
* Patient showing either postprandial fullness, bloating in the upper abdomen, or early satiation as the major complaint among the 8 symptoms shown below at the time of obtaining consent

  * upper abdominal pain
  * upper abdominal discomfort
  * postprandial fullness
  * bloating in the upper abdomen
  * early satiation
  * nausea
  * vomiting
  * belching
* Outpatient

Exclusion Criteria:

* Patient showing symptoms of organic disease (reflux esophagitis, erosion, ulceration, esophageal hiatal hernia, bleeding, malignant tumor, Barrett's esophagus) when upper gastrointestinal endoscopy is performed within 24 weeks before obtaining consent
* Patient showing heartburn within 12 weeks before obtaining consent
* Patient complicated by irritable bowel syndrome
* Patient complicated by diabetes mellitus requiring medication
* Patient complicated by severe anxiety disorder with some problems in interpersonal relationships or social life
* Patient complicated by depression (including suspected cases) or sleep disturbance

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2008-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Subject's global assessment | Every week

SECONDARY OUTCOMES:
Disappearance rate of symptoms | Every week
Laboratory tests, resting | At 0, 4, 12, 24, 36, 48 week
12-lead ECG | At 0, 24 and 48 week
Adverse events | During treatment

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Inc
Locations (4):
- Japan (4):
  - Hokkaido
  - Kansai
  - Kantou
  - Kyushu

REFERENCES:
- [Background] Matsueda K, Hongo M, Ushijima S, Akiho H. A long-term study of acotiamide in patients with functional dyspepsia: results from an open-label phase III trial in Japan on efficacy, safety and pattern of administration. Digestion. 2011;84(4):261-8. doi: 10.1159/000332404. Epub 2011 Sep 21. PMID 21934307